CLINICAL TRIAL: NCT03480217
Title: Assessing the Effectiveness of a Multifaceted Implementation Strategy to Increase the Uptake of the USPSTF Hypertension Screening Recommendations in an Ambulatory Care Network: a Cluster Randomized Trial
Brief Title: Implementing Hypertension Screening Guidelines in Primary Care
Acronym: EMBRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Ian Kronish, Florence Irving Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAQ1062; 1R01HS024262-01 (AHRQ)
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Hypertension,Essential; White Coat Hypertension
Keywords: hypertension; screening; guidelines; implementation; randomized
MeSH Terms: conditions — Essential Hypertension; White Coat Hypertension; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to group assignment when coding medical records to determine whether providers ordered out-of-office BP testing for eligible patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Clinics, Pre-Implementation (Experimental): Usual care
  Interventions: Other: Usual care
- Intervention Clinics, Post-Implementation (Experimental): Patients will be screened for hypertension by primary care clinicians, registered nurses, medical assistants, and front desk staff from clinics randomized to receive the Multifaceted Implementation Strategy.
  Interventions: Behavioral: Multifaceted Implementation Strategy
- Control Clinics, Pre-Implementation (Other): Usual care
  Interventions: Other: Usual care
- Control Clinics, Post-Implementation (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Multifaceted Implementation Strategy — Key components include:
  * educational presentations to primary care providers at grand rounds
  * patient information materials on ABPM and HBPM
  * training registered nurses to assist providers with teaching patients to conduct HBPM
  * information on how to order ABPM and HBPM to clinicians, nurses and front desk staff via huddles, emails, and other electronic communications
  * a computerized EHR-embedded clinical decision support tool that prompts providers to recall the USPSTF hypertension guidelines and facilitates ordering of HBPM and ABPM for guideline-eligible patients
  * periodic feedback to primary care providers about clinic-level success with appropriately ordering ABPM and HBPM for eligible patients
  * an accessible, culturally-adapted and locally tailored ABPM service
  Arms: Intervention Clinics, Post-Implementation
Other: Usual care — Primary care clinicians diagnose hypertension according to usual care
  Arms: Control Clinics, Post-Implementation; Control Clinics, Pre-Implementation; Intervention Clinics, Pre-Implementation

SUMMARY:
The goal of this study is to use a cluster-randomized design (1:1 ratio) among 8 primary care clinics affiliated with New York-Presbyterian Hospital to test the effectiveness of a theory-informed multifaceted implementation strategy designed to increase the uptake of the 2015 United States Preventive Services Task Force (USPSTF) hypertension screening guidelines. The primary outcome is the ordering of out-of-office blood pressure testing, either ambulatory blood pressure monitoring (ABPM) or home blood pressure monitoring (HBPM), by primary care clinicians for patients with newly elevated office blood pressure (BP), as recommended by the 2015 guidelines.

DETAILED DESCRIPTION:
The goal of this study is to assess the effect of a multifaceted implementation strategy aimed at increasing adherence to the 2015 U.S. Preventive Services Task Force (USPSTF) recommendations for hypertension screening, with a focus on implementation in primary care clinics that reach medically underserved patients. The accurate diagnosis of hypertension is essential for targeting appropriate therapy at the patients who can most benefit from hypertension treatment. On the other hand, inappropriate diagnosis of hypertension can lead to unnecessary treatment with blood pressure (BP) medications, wasteful healthcare utilization, and adverse psychological consequences from being mislabeled as having a chronic disease.

There are challenges to measuring BP in clinical settings that make inappropriate diagnosis common. A systematic review conducted by the USPSTF in 2014 found that 5%-65% of patients with elevated office BP do not have high out-of-office BP readings according to ambulatory BP monitoring (ABPM) or home BP monitoring (HBPM). This is commonly referred to as white-coat hypertension. In contrast to patients with sustained hypertension (elevated BP in office and out-of-office settings), patients with white-coat hypertension do not appear to be at increased cardiovascular risk nor to benefit from antihypertensive treatment. Based primarily on these observations, in 2015, the USPSTF updated their hypertension screening guidelines to recommend that patients with elevated office BP undergo out-of-office BP testing (ABPM or HBPM) to rule-out white-coat hypertension prior to a new diagnosis of hypertension. While ABPM is recommended as the first-line out-of-office screening test, HBPM is cited as a reasonable alternative if ABPM is unavailable.

Despite the USPSTF guideline recommendation, ABPM and HBPM are currently infrequently utilized in the US, particularly as part of hypertension diagnosis. Accordingly, the investigators conducted focus groups with primary care providers, patients, and other key stakeholders (medical directors, nurse supervisors, medical assistants, nurse practitioners, front desk staff) to identify the major barriers to implementation of the new hypertension screening guidelines. The investigators then applied the Behavior Change Wheel, a trans-theoretical intervention development framework, to categorize barriers and select theory-informed intervention components that would address these barriers. The investigators arrived at a theory-informed implementation strategy for improving out-of-office BP testing, which included educational activities for providers (i.e., presentations at grand rounds or other venues at which physicians are present); training registered nurses to be capable of assisting with teaching patients to conduct HBPM; disseminating information on how to order ABPM and HBPM to clinicians, nurses, and front desk staff via huddles, emails, and other electronic communications; creating a computerized electronic health record (EHR)-embedded clinical decision support tool that prompts recall of the USPSTF hypertension guidelines and facilitates ordering of HBPM and ABPM for eligible patients; creating and disseminating patient information materials on ABPM and HBPM; providing periodic feedback about clinic-level success with adhering to the guideline, and developing an easily accessible, culturally-adapted and locally tailored ABPM service.

The investigators now aim to test this multifaceted implementation strategy to increase the uptake of the USPSTF hypertension recommendations in the ambulatory care network (ACN) of New York-Presbyterian Hospital (NYP), a network of primary care clinics serving 120,000 patients from underserved communities in New York City. Specifically, the investigators are conducting a 2-year cluster randomized trial (Phase II of the project) following a 6-month implementation phase in which we randomize matched pairs of 8 ACN clinics (1:1) to either receive the multicomponent guideline implementation strategy (N = 4 clinics) or a wait-list control (N = 4 clinics). The investigators aim to assess the effectiveness of this intervention on the completion of out-of-office BP testing (ABPM or HBPM) prior to hypertension diagnosis (primary outcome) as well as the effect on out-of-office test ordering, irrespective of test completion (secondary outcome).

ELIGIBILITY:
Patient Inclusion Criteria (as per electronic medical records):

* Elevated blood pressure (BP) (systolic BP>=140 mmHg or diastolic BP >=90 mmHg) at a scheduled clinic visit with a primary care provider from a clinic that is participating in the study; if multiple BP readings were taken from a visit, then the average of the readings will be used

Patient Exclusion Criteria (as per electronic medical records):

* Prior diagnosis of hypertension
* Prior diagnosis of white-coat hypertension
* Prior evaluation for white-coat hypertension by 24-hr ABPM or HBPM
* Prescribed antihypertensive medication
* Manual office BP <140/90 mmHg
* Severely elevated BP (systolic BP>=180 mmHg or diastolic BP>=110 mmHg)
* Evidence of target-organ damage (chronic kidney disease, cardiovascular disease)

Clinic Inclusion Criteria:

* Primary care clinics that are part of the New York-Presbyterian Hospital Ambulatory Care Network and were not part of implementation development

Clinic Exclusion Criteria:

* Medical director of clinic declines to participate in cluster randomized trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kronish, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Center for Behavioral Cardiovascular Health, New York, New York
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data archive that contains raw study data will be posted on an open science platform.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 1 year of completion of study activities
Access Criteria: Access to the data archive will be provided upon request.

REFERENCES:
- [Background] Siu AL; U.S. Preventive Services Task Force. Screening for high blood pressure in adults: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2015 Nov 17;163(10):778-86. doi: 10.7326/M15-2223. Epub 2015 Oct 13. PMID 26458123
- [Background] Kronish IM, Kent S, Moise N, Shimbo D, Safford MM, Kynerd RE, O'Beirne R, Sullivan A, Muntner P. Barriers to conducting ambulatory and home blood pressure monitoring during hypertension screening in the United States. J Am Soc Hypertens. 2017 Sep;11(9):573-580. doi: 10.1016/j.jash.2017.06.012. Epub 2017 Jul 6. PMID 28734798
- [Background] Piper MA, Evans CV, Burda BU, Margolis KL, O'Connor E, Whitlock EP. Diagnostic and predictive accuracy of blood pressure screening methods with consideration of rescreening intervals: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2015 Feb 3;162(3):192-204. doi: 10.7326/M14-1539. PMID 25531400
- [Background] Moise N, Phillips E, Carter E, Alcantara C, Julian J, Thanataveerat A, Schwartz JE, Ye S, Duran A, Shimbo D, Kronish IM. Design and study protocol for a cluster randomized trial of a multi-faceted implementation strategy to increase the uptake of the USPSTF hypertension screening recommendations: the EMBRACE study. Implement Sci. 2020 Aug 8;15(1):63. doi: 10.1186/s13012-020-01017-8. PMID 32771002
- [Background] Carter EJ, Moise N, Alcantara C, Sullivan AM, Kronish IM. Patient Barriers and Facilitators to Ambulatory and Home Blood Pressure Monitoring: A Qualitative Study. Am J Hypertens. 2018 Jul 16;31(8):919-927. doi: 10.1093/ajh/hpy062. PMID 29788130
- [Result] Kronish IM, Phillips E, Alcantara C, Carter E, Schwartz JE, Shimbo D, Serafini M, Boyd R, Chang M, Wang X, Razon D, Patel A, Moise N. A Multifaceted Implementation Strategy to Increase Out-of-Office Blood Pressure Monitoring: The EMBRACE Cluster Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2334646. doi: 10.1001/jamanetworkopen.2023.34646. PMID 37747734
- [Derived] Kronish IM, Carter E, Phillips E, Alcantara C, Serafini M, Schwartz JE, Moise N. Impact of a Theory-Informed Implementation Strategy on Clinician Attitudes Toward Out-of-Office Blood Pressure Monitoring for Hypertension Screening. J Gen Intern Med. 2025 Oct 14. doi: 10.1007/s11606-025-09840-9. Online ahead of print. PMID 41085961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were passively recruited from the electronic health record.
Pre-assignment Details: This 2-group, pre-post cluster randomized trial was conducted within a primary care network of 8 practices and 1186 patients (857 intervention; 329 control). Depending on the practice/clinic and the implementation period, patients will receive usual care or care that has been impacted by the multifaceted implementation strategy.
Units Other Than Participants: clinics
Groups:
- Intervention Clinics: Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to receive the implementation strategy before the multifaceted implementation strategy had been delivered (i.e., pre-implementation period, no exposure to intervention)
- Control (Usual Care) Clinics: Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to not receive the multifaceted implementation strategy and receive usual care before the implementation period begins (i.e., pre-implementation period, no exposure to intervention)
Period: Pre-Implementation (12 Months)
Arm/Group | Intervention Clinics | Control (Usual Care) Clinics
Started | 456; 8 clinics | 139; 8 clinics
Completed | 456; 8 clinics | 139; 8 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics
Period: Post-Implementation (12 Months)
Arm/Group | Intervention Clinics | Control (Usual Care) Clinics
Started | 401; 8 clinics | 190; 8 clinics
Completed | 401; 8 clinics | 190; 8 clinics
Not Completed | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Population: The clinics are either implementing the intervention (4 out of 8) or providing usual care (4 out of 8) after the implementation period begins. The baseline analysis for the participants that visited these clinics are calculated separately - those who visited the Intervention Clinics before and after the implementation (456+401=857 total) and those who visited the Control Clinics before and after the implementation (139+190=329 total).
Groups:
- Intervention Clinics (Pre-Implementation): Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to receive the implementation strategy before the multifaceted implementation strategy had been delivered (i.e., pre-implementation period, no exposure to intervention)
- Intervention Clinics (Post-Implementation): Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to receive the implementation strategy after the multifaceted implementation strategy had been delivered (i.e., post-implementation period, exposure to intervention)
- Control (Usual Care) Clinics (Pre-Implementation): Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to not receive the multifaceted implementation strategy and receive usual care before the implementation period begins (i.e., pre-implementation period, no exposure to intervention)
- Control (Usual Care) Clinics (Post-Implementation): Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to not receive the multifaceted implementation strategy and receive usual care after the implementation period begins (i.e., post-implementation period, no exposure to intervention)
- Total: Total of all reporting groups
Arm/Group | Intervention Clinics (Pre-Implementation) | Intervention Clinics (Post-Implementation) | Control (Usual Care) Clinics (Pre-Implementation) | Control (Usual Care) Clinics (Post-Implementation) | Total
Number analyzed (Participants) | 456 | 401 | 139 | 190 | 1186
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.1) | 51.3 (14.5) | 58.9 (16.0) | 59.8 (19.1) | 53.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 257 | 105 | 157 | 808
  Male | 167 | 144 | 34 | 33 | 378
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 152 | 113 | 50 | 53 | 368
  Not Hispanic or Latino | 70 | 79 | 17 | 43 | 209
  Unknown or Not Reported | 234 | 209 | 72 | 94 | 609
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 53 | 50 | 9 | 11 | 123
  White | 86 | 69 | 33 | 57 | 245
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 317 | 282 | 97 | 122 | 818
Region of Enrollment [Number; unit: participants]
  United States | 456 | 401 | 139 | 190 | 1186

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patient Visits With Completion of Out-of-office BP Monitoring Within 6 Months of an Eligible Visit During the Pre-Implementation Period
Description: Patient completed out-of-office BP testing [ambulatory blood pressure monitoring (ABPM) or home blood pressure monitoring (HBPM)] (either Y/N) per eligible visits were tallied.
Time Frame: 6 months (Pre-Implementation period)
Measure: Number; unit: percentage of visits
Units Other Than Participants: number of visits
Groups:
- Intervention Clinics: Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to receive the implementation strategy.
  Patients receive usual care if they come before the implementation period (pre-implementation period) and receive care that has been impacted by the multifaceted implementation strategy if they attend visits after the implementation period (post-implementation period).
- Control Clinics: Participants are patients with elevated office blood pressure and no prior diagnosis of hypertension who attend primary care visits at clinics that were randomly allocated to receive usual care.
  Patients receive usual care if they come before the implementation period (pre-implementation period) and receive usual care if they attend visits after the implementation period (post-implementation period).
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | 456 | 139
Number analyzed (number of visits) | 529 | 149
percentage of visits | 0.6 | 5.4

2. Secondary Outcome: Percentage of Patient Visits With Out-of-office BP Monitoring Test Ordered by Clinician During the Pre-Implementation Period
Description: Primary care clinician ordered out-of-office BP testing [ABPM or HBPM] (either Y/N) for eligible visits were tallied.
Time Frame: 6 months (Pre-Implementation period)
Measure: Number; unit: percentage of visits
Units Other Than Participants: number of visits
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | 456 | 139
Number analyzed (number of visits) | 529 | 149
percentage of visits | 2.8 | 8.7

3. Primary Outcome: Percentage of Patient Visits With Completion of Out-of-office BP Monitoring Within 6 Months of an Eligible Visit During the Post-Implementation Period
Description: as for outcome 1
Time Frame: 6 months (Post-Implementation period)
Measure: Number; unit: percentage of visits
Units Other Than Participants: number of visits
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | 401 | 190
Number analyzed (number of visits) | 454 | 207
percentage of visits | 5.7 | 4.3

4. Secondary Outcome: Percentage of Patient Visits With Out-of-office BP Monitoring Test Ordered by Clinician During the Post-Implementation Period
Description: Primary care clinician ordered out-of-office BP testing [ABPM or HBPM] (either Y/N) for eligible visits were tallied.
Time Frame: 6 months (Post-Implementation period)
Measure: Number; unit: percentage of visits
Units Other Than Participants: number of visits
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | 401 | 190
Number analyzed (number of visits) | 454 | 207
percentage of visits | 7.9 | 9.2

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded up to 6 months after the 12-month pre-implementation and 12-month post-implementation periods.
Description: Adverse events related to ABPM testing were reported in the Columbia ABPM testing service clinical database. Other adverse events were collected if reported in the electronic health record.
Arm/Group | Intervention Clinics | Control Clinics
All-Cause Mortality (participants affected / at risk) | 0/857 | 0/329
Serious Adverse Events (participants affected / at risk) | 0/857 | 0/329
Other Adverse Events (participants affected / at risk) | 0/857 | 0/329

LIMITATIONS AND CAVEATS:
The Coronavirus Disease 2019 (COVID-19) pandemic led to the closure of the ABPM testing service during the maintenance period which precluded an evaluation of the implementation strategy during the maintenance period. Additionally, a new electronic health record was adopted in 2020 which also precluded an evaluation of the use of HBPM during the maintenance period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03480217/Prot_SAP_000.pdf